CLINICAL TRIAL: NCT06162611
Title: Generating Evidence to Improve Same-day Etonogestrel (ENG) Implant Insertion for Emergency Contraception
Brief Title: Etonogestrel (ENG) Implant Insertion for Emergency Contraception With Oral Levonorgestrel (LNG) vs Placebo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lori Gawron (Other)
Collaborators: Planned Parenthood Association of Utah (Unknown)
Responsible Party: Sponsor-Investigator, Lori Gawron, Associate Professor OBGYN, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00152448
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Emergency Contraception
Keywords: contraception; etonogestrel implant; oral levonorgestrel
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of the etonogestrel contraceptive implant randomized to same day oral levonorgestrel or placebo in emergency contraception patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The University of Utah Investigational Pharmacy encapsulated oral levonorgestrel and placebo pills and applied a randomization scheme that will not be broken until end of study or at the request of the data safety monitoring board
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Etonogestrel contraceptive implant with oral levonorgestrel (Active Comparator): Patients will be randomized 1:1 to each arm and will receive the contraceptive implant with a same-day encapsulated pill with either oral levonorgestrel 1.5mg
  Interventions: Drug: Etonogestrel implant with Oral Levonorgestrel emergency contraception 1.5mg
- Etonogestrel contraceptive implant with placebo (Placebo Comparator): Patients will be randomized 1:1 to each arm and will receive the contraceptive implant with a same-day encapsulated pill with placebo X 1 dose
  Interventions: Device: Etonogestrel implant with oral placebo

INTERVENTIONS:
Drug: Etonogestrel implant with Oral Levonorgestrel emergency contraception 1.5mg — Single pill of oral levonorgestrel 1.5mg X 1 dose (e.g. Plan B) same day as contraceptive implant insertion
  Arms: Etonogestrel contraceptive implant with oral levonorgestrel
Device: Etonogestrel implant with oral placebo — Single pill of placebo same day as contraceptive implant insertion
  Arms: Etonogestrel contraceptive implant with placebo

SUMMARY:
Intrauterine devices (IUDs) are highly effective to prevent pregnancy when used for emergency contraception (following unprotected intercourse in the last 3 days), but data are lacking for people who desire an etonogestrel (ENG) contraceptive implant in this situation. This proposal will identify the most effective way to start an implant for emergency contraception using a randomized controlled trial comparing pregnancy risk between those receiving the implant vs. the implant plus oral emergency contraception (EC). Data from this project will inform clinical practice and add another option, the implant, for those desiring a long acting, highly effective contraceptive method when they present for emergency contraception.

DETAILED DESCRIPTION:
Oral emergency contraception (EC), is commonly used after recent unprotected intercourse to avoid undesired pregnancy, but does not provide ongoing contraception. Rigorous data allow for use of intrauterine devices (IUDs) as both EC and ongoing contraception, but EC efficacy data on use of the etonogestrel (ENG) implant, is lacking. The CDC Selected Practice Recommendations for Contraceptive Use support initiation of the ENG implant if oral levonorgestrel (LNG) is given concomitantly for EC. This recommendation lacks supporting evidence and serves as a barrier to method initiation, as oral LNG is not typically available in clinics when clients desire an implant. Additionally, oral LNG efficacy decreases in higher body mass index (BMI) users and the role of BMI on efficacy with co-administered oral LNG and the ENG implant is unknown. As the ENG implant is also a synthetic progestogen with a rapid rise and consistent systemic levels, it could plausibly serve as stand-alone EC or increase the efficacy of oral LNG with co-administration. Moreover, the EC mechanism of action, which is related to ovulatory suppression with oral EC, may differ if the implant is initiated with or without oral LNG, impacting efficacy in mid cycle users. This study addresses the following research gaps around use of the ENG implant for EC that serve as barriers to provider comfort with these options: efficacy with and without oral LNG, efficacy differences by BMI, and ovulation frequency with and without oral LNG. The investigators propose a randomized, placebo-controlled, non-inferiority study to determine if the ENG implant alone is no worse than the ENG implant + oral LNG for EC, using a 3.5% non-inferiority margin. The investigators will include clients who present to Planned Parenthood Association of Utah clinics with report of unprotected intercourse within 72 hours who desire EC. Eligible EC clients interested in an implant with a negative pregnancy test will be allocated 1:1 to a study group: (1) ENG implant + oral LNG or (2) ENG implant + placebo. Our experienced research staff will follow up with participants for 4-week efficacy data as primary outcome. Our aims include: (1) To compare the efficacy of the ENG Implant + oral LNG to the ENG Implant + placebo for EC in 790 participants assessed by pregnancy status four weeks after implant placement, (2) To compare pregnancy risk by BMI category (the investigators anticipate half of the 790 participants will have a BMI ≥25) between and within the ENG Implant + oral LNG and the ENG Implant + placebo groups, and (3) To evaluate ovulation frequency within 5 days of insertion of ENG Implant + oral LNG or ENG implant + placebo in 202 participants who are mid cycle (day 7-14 post menses) at time of enrollment assessed by serum progesterone levels and urine fertility monitor results. Our short-term goal is to expand evidence on the efficacy of implant initiation with or without oral LNG to meet the needs of EC clients. Our long-term goals are to develop evidence-based clinical guidelines to inform global contraceptive practices, allow for equity in long acting reversible contraception counseling at the time of EC, and support reproductive autonomy for people to achieve to their life goals.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-35 years old
* Unprotected intercourse within 72 hours
* Biologically capable of pregnancy (intact uterus without prior sterilization surgery
* Fluent in English and/or Spanish
* Have a regular menstrual cycle (21-35 days)
* Known last menstrual period (+/- 3 days)
* Working (cell) phone number
* Willing to comply with the study requirements
* Willing to abstain from any CYP3A4 inducer for 5 days

Exclusion Criteria:

* Current pregnancy (+urine pregnancy test in clinic)
* Breastfeeding
* Contraindication to ENG or LNG based on CDC MEC/SPR
* Sterilization, hysterectomy, or has an IUD or contraceptive implant in place
* Vaginal bleeding of unknown etiology
* Previous use of EC in same cycle
* Allergy to LNG or ENG
* History of intolerance/ side effects with ENG Implant
* Current (past 7 days) use of any CYP3A4 inducer
* Plan to use any other steroid hormone in the next 4 weeks (testosterone, estrogen, progesterone)
* Ended a pregnancy at or under 20 weeks gestational age within last 2 weeks
* Ended a pregnancy over 20 weeks gestational age in last 6 weeks
* Use of any injectable hormonal contraceptive (Depo-Provera) in the last 15 weeks
* Use of any oral EC, contraceptive pills, patches, vaginal rings, or an IUD or Implant in the last 2 weeks

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 790 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the etonogestrel contraceptive implant with placebo for emergency contraception | 1 month after enrollment
  Pregnancy rate = number of pregnancies / participants in the placebo arm
Efficacy of the etonogestrel contraceptive implant with placebo for emergency contraception by BMI category | 1 month after enrollment
  Pregnancy rate = # of pregnancies / participants in the placebo arm stratified by BMI category
Efficacy of the etonogestrel contraceptive implant with oral levonorgestrel for emergency contraception | 1 month after enrollment
  Pregnancy rate = # of pregnancies / participants in the oral levonorgestrel arm
Efficacy of the etonogestrel contraceptive implant with oral levonorgestrel for emergency contraception by BMI category | 1 month after enrollment
  Pregnancy rate = # of pregnancies / participants in the oral levonorgestrel arm stratified by BMI category
Ovulation frequency within 5 days of implant insertion in the oral levonorgestrel arm | 5 days after implant insertion
  Incidence of ovulation within 5 days after implant insertion measured by urine fertility monitor results and serum progesterone
Ovulation frequency within 5 days of implant insertion in the placebo arm | 5 days after implant insertion
  Incidence of ovulation within 5 days after implant insertion measured by urine fertility monitor results and serum progesterone

SECONDARY OUTCOMES:
Implant continuation | 4 weeks after insertion
  Participants continuing implant use at one month as a proportion of all participants having successful placement of implant at study entry. Measured by probabilities estimated using Kaplan-Meier approach.
Implant satisfaction | 4 weeks after insertion
  Likelihood of satisfaction by study group using ordinal regression. Measured by 5-point ordinal scale (5-point ordinal scale: (1) very unsatisfied, (2) unsatisfied, (3) neutral, (4) satisfied, (5) very satisfied). Measured by

CONTACTS AND LOCATIONS:
Overall Officials: Lori Gawron, MD, MPH, Principal Investigator — University of Utah
Locations (1):
- Planned Parenthood Association of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No